CLINICAL TRIAL: NCT04965311
Title: A Phase II Trial of Pre-Operative Endoscopic Botulinum Toxin Injection in the Prevention of Postoperative Pancreatic Fistula Following Distal Pancreatectomy
Brief Title: Endoscopic Botulinum Toxin Injection in the Prevention of Postoperative Pancreatic Fistula Following Distal Pancreatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brett C. Sheppard, M.D., FACS, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022619; NCI-2021-06239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022619 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA; prabotulinumtoxin A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment of POPF (botulinum toxin type A) (Experimental): Patients receive botulinum toxin type A via endoscopic injection into intraduodenal sphincter of Oddi segment between 7-14 days prior to planned distal pancreas resection.
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Given via endoscopic injection into intraduodenal sphincter of Oddi segment
  Other Names: AbobotulinumtoxinA; Botox; Botox Cosmetic; Botulinum A Toxin; Botulinum Neurotoxin Type A; Botulinum Toxin A; BTX-A; DaxibotulinumtoxinA; Dysport; EvabotulinumtoxinA; IncobotulinumtoxinA; OnabotulinumtoxinA; Onaclostox; Prabotulinumtoxin A; Xeomin

SUMMARY:
This phase II trial studies the effect of botulinum toxin (Botox) in preventing postoperative pancreatic fistula after distal pancreatectomy. Postoperative pancreatic fistula (POPF) is a known risk of distal pancreatic surgery, in which leakage of pancreatic digestive liquids causes internal swelling that can be painful (termed inflammation). A valve-like muscle, called the Sphincter of Oddi, opens and closes, controlling the flow of digestive liquids from the liver (bile) and pancreas (pancreatic juice) to the small intestine (duodenum). After surgery, the Sphincter of Oddi may act to block the flow of normal pancreatic secretions, causing secretions to leak into the abdomen resulting in POPF. Botox is a drug that can cause paralysis of muscles. Giving an injection of Botox into the sphincter of Oddi before distal pancreatic surgery may reduce leakage of digestive fluids and potential POPF.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of pre-operative botulinum toxin type A (BTX) injection compared to no therapy for the prevention of clinically relevant POPF.

SECONDARY OBJECTIVES:

I. Evaluate the safety of pre-operative BTX injection into the Sphincter of Oddi.

II. Evaluate the efficacy of pre-operative BTX injection compared to no therapy for the prevention of all POPF.

EXPLORATORY OBJECTIVES:

I. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in POPF.

II. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in clinically relevant POPF (crPOPF).

III. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in postoperative length of hospital stay.

IV. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in rate of Clavien-Dindo grade III or greater complications.

V. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in rate of percutaneous drainage.

VI. Using a historical population matched for potential confounding clinicopathologic variables, evaluate differences in rate of unplanned re-operation.

OUTLINE:

Patients receive botulinum toxin type A via endoscopic injection into intraduodenal sphincter of Oddi segment between 7-14 days prior to planned distal pancreas resection.

Patients are followed for 30 days following distal pancreas resection.

ELIGIBILITY:
Inclusion Criteria:

* Participant scheduled for elective distal pancreatectomy or radical antegrade modular pancreatosplenectomy (RAMPS), via open or laparoscopic technique
* Participant >= 18 years of age
* Ability to understand nature and individual consequences of clinical trial
* Written informed consent from participant or legally authorized representative
* For participants of childbearing potential, a negative pregnancy test and adequate contraception until 14 days after trial intervention

Exclusion Criteria:

* Known hypersensitivity to any BTX preparation or to any of the components in the formulation
* Infection at the proposed injection site, including cholangitis
* Anatomy incompatible with planned intervention (e.g., Roux-en-Y gastric bypass, distal gastrectomy with Roux-en-Y or Billroth II reconstruction)
* Acute pancreatitis within 2 weeks of planned study intervention
* American Society of Anesthesiologists (ASA) score > III
* Serious cardiovascular disease (e.g., myocardial infarction in the past year, New York Heart Association [NYHA] III/IV congestive heart failure, unstable angina)
* Creatinine clearance < 30 mL/min
* Liver cirrhosis (of any Child-Pugh grade)
* Neuromuscular or any neurological disease with associated increased risk for a participant undergoing BTX injection
* Prior BTX administration
* Inability to obtain informed consent due to comprehension or language barrier
* Inability to comply with study and/or follow-up procedures
* Pregnancy or lactation
* Any condition that could result in undue risk for the participant and/or influence outcome measures (in the opinion of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett C Sheppard, M.D., FACS, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 58.75 [50 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Relevant Postoperative Pancreatic Fistula (POPF)
Description: Defined by standard biochemical definitions of POPF per the International Study Group of Pancreatic Fistula (ISGPF) criteria.
Time Frame: Up to postoperative day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Rate of Serious Adverse Event
Description: Using the safety analysis set, the rate of serious adverse events following endoscopic BTX injection into the sphincter of Oddi as a single agent will be determined for participants undergoing distal pancreas resections. The 95% confidence interval will be reported with the point estimate of serious adverse events (SAE) rate.
Time Frame: Prior to surgery up to 30 days post surgery (up to 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
Number analyzed (Participants) | 4
Participants | 1

3. Secondary Outcome: Number of Participants With Any POPF
Time Frame: Prior to surgery up to 30 days post surgery (up to 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Prior to surgery up to 30 days post surgery
Arm/Group | Treatment of POPF (Botulinum Toxin Type A)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment of POPF (Botulinum Toxin Type A) (N=4)
Inpatient Hospitalization (Renal and urinary disorders) | 1 (1) — Patient was re-admitted to the hospital on 4/5/2023 after follow-up clinic labs demonstrated acute AKI. SAE assessed as unrelated to study participation but rather a surgical technical error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT04965311/Prot_SAP_000.pdf